CLINICAL TRIAL: NCT00631865
Title: Autologous Transplantation of Melanocytes for Treatment of Vitiligo Skin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-skin-001
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2009-02

CONDITIONS: Vitiligo
Keywords: melanocytes
MeSH Terms: conditions — Vitiligo | interventions — Cell- and Tissue-Based Therapy; Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cell transplantation group (Experimental): Epidermal Cell transplantation in patients with vitiligo
  Interventions: Biological: Melanocyte transplantation

INTERVENTIONS:
Biological: Melanocyte transplantation — Injection of melanocytes directly in Epidermis
  Other Names: cell therapy; cell transplantation

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of melanocytes in patients with vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a pigmentation disorder in which white patches of skin appear on different parts of the body. Histologically it is characterized by absence of melanocytes along the epidermal basal layer.

Using cell suspension with non-cultured melanocytes which injected into blister of depigmented lesion, a success rate of 85% was reported for repigmentation. However there are some limitations in this technique: the induction of blister is limited to several sites of the body, hypo-pigmentation around the recipient area due to cryodamage of peripheral melanocytes and leakage of suspension out of the blister. To reduce these problems, in this study we will inject melanocytes directly to epidermis.

A shaved biopsy specimen (about 1 cm2) is taken from the patient's normally pigmented area under local anesthesia (lidocaine hydrochloride 20 mg/ml). The specimens are incubated in 0.25% trypsin solution for 15 minutes at 37°C 0.02% EDTA solution for 10 minutes. Then epidermal sheets are gently manipulated with forceps to dissociate the epidermal cells and to yield a cell suspension, followed by treatment with 0.5% trypsin/versene solution at 37C for 3-5 minutes. Well-dispersed cell suspension is aspirated into 1 ml syringes and injected directly in epidermis.

ELIGIBILITY:
Inclusion Criteria:

* Age over 12 years
* Stable form of vitiligo (no increase in the size of the lesion for at least one year)
* No use of immunosuppressive & cytotoxic drugs at least for past 6 months

Exclusion Criteria:

* Pregnant patients
* Patients with active disease
* Infection at the recipient site
* Evidence of köebner in the past
* Keloidal tendencies

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-02; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
percentage of repigmentation | 2 and 4 weeks after transplantation

SECONDARY OUTCOMES:
stability of the achieved repigmentation | 6 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Baharvand, PhD, Principal Investigator — Head of Royan stem cell department; Saeeid Shafieian, MD, Principal Investigator — Firoozgar Hospital; Nasser Aghdami, MD., PhD, Study Director — Head of Royan transplantation Lab
Locations (1):
- Royan Institute, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Khodadadi L, Shafieyan S, Sotoudeh M, Dizaj AV, Shahverdi A, Aghdami N, Baharvand H. Intraepidermal injection of dissociated epidermal cell suspension improves vitiligo. Arch Dermatol Res. 2010 Oct;302(8):593-9. doi: 10.1007/s00403-010-1034-7. Epub 2010 Apr 4. PMID 20364383
- See also: Related Info — http://www.royaninstitute.org